CLINICAL TRIAL: NCT01282762
Title: An Observational Study Evaluating the Long-Term Safety and Immunogenicity of HEPLISAV™ Compared With Engerix-B® in Adults With Chronic Kidney Disease Who Have Previously Received At Least One Hepatitis B Vaccine Series
Brief Title: Long-Term Study on Safety and Immunogenicity of HEPLISAV™ and Engerix-B® in Adults With Chronic Kidney Disease
Status: Completed | Type: Observational
Sponsor: Dynavax Technologies Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: DV2-HBV-19
Record Dates: First submitted 2011-01-20; First posted 2011-01-25 (Estimated); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Chronic Kidney Disease
Keywords: Prevention of Hepatitis B infection.; End Stage Renal Disease; Hepatitis B vaccination; Hepatitis B virus (HBV)
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic; Hepatitis B | interventions — Hepatitis B Vaccines; Engerix-B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum retained during study duration for additional testing if indicated
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: HEPLISAV — 0.5 mL administered intramuscularly (IM) at Week 0, Week 4 and Week 24.
  HEPLISAV booster injection = one dose of 0.5 mL volume when needed.
  Other Names: Hepatitis B vaccine (recombinant), adjuvanted
Biological: Engerix-B — 2.0 mL administered intramuscularly (IM) at Week 0, Week 4, Week 8 and Week 24.
  Engerix-B booster injection = one dose of 2.0 mL volume when needed
  Other Names: Hepatitis B vaccine (recombinant)

SUMMARY:
The purpose of this study is to determine the durability of seroprotection of HEPLISAV™ and Engerix-B® and the number of injections of each vaccine needed to maintain seroprotection in a cohort of chronic kidney disease (CKD) patients over time.

DETAILED DESCRIPTION:
An Observational Study Evaluating the Long-Term Safety and Immunogenicity of HEPLISAV™ compared with Engerix-B® in Adults with Chronic Kidney Disease who Have Previously Received At Least One Hepatitis B Vaccine Series

ELIGIBILITY:
Inclusion Criteria:

A subject must meet all of the following inclusion criteria to participate in the study:

* enrolled and completed HEPLISAV or Engerix-B treatment in: DV2-HBV-17 or DV2-HBV-18 and had anti-HBsAg ≥ 10 mIU/mL prior to or during DV2-HBV-18
* previously received a complete primary hepatitis B vaccine series in DV2-HBV-17 or prior to enrollment in DV2-HBV-18
* be otherwise clinically stable in the opinion of the investigator
* be able and willing to provide informed consent

Exclusion Criteria:

A subject who meets any ONE of the following exclusion criteria is not permitted to participate in the study:

* previously enrolled in DV2-HBV-18 and never obtained anti-HBsAg ≥ 10 mIU/mL
* received hepatitis B vaccine off-study after enrolling in DV2-HBV-17 or DV2-HBV-18
* has known history of autoimmune disease
* is unwilling or unable to comply with all the requirements of the protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with Chronic Kidney Disease previously enrolled in the Dynavax clinical studies DV2-HBV-17 and DV2-HBV-18
Sampling Method: Non-Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2010-12; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the durability of seroprotection induced by HEPLISAV and Engerix-B as measured by seroprotection rate (SPR) (anti-HBsAg> 10 milli-international unit (mIU)/mL | Baseline
To evaluate the durability of seroprotection induced by HEPLISAV and Engerix-B as measured by SPR (anti-HBsAg> 10 mIU/mL | 6 months
To evaluate the durability of seroprotection induced by HEPLISAV and Engerix-B as measured by SPR (anti-HBsAg> 10 mIU/mL | 12 months
To evaluate the durability of seroprotection induced by HEPLISAV and Engerix-B as measured by SPR (anti-HBsAg> 10 mIU/mL | 24 months
To evaluate the durability of seroprotection induced by HEPLISAV and Engerix-B as measured by SPR (anti-HBsAg> 10 mIU/mL | 36 months
To evaluate the durability of seroprotection induced by HEPLISAV and Engerix-B as measured by SPR (anti-HBsAg> 10 mIU/mL | 48 months

SECONDARY OUTCOMES:
To evaluate the safety of HEPLISAV and Engerix-B in CKD subjects who previously received at least one hepatitis B vaccine series. | Baseline and 6,12, 24, 36 and 48 months

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Associates of Tidewater, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided
No Changes to status a/o 3/2017

REFERENCES:
- [Derived] Girndt M, Houser P, Manllo-Karim R, Ervin JE, Charytan C, Chow S, Symonian-Silver M, Lehrner L, Linfert D, Shemin D, Michelsen A, Xie F, Janssen RS. Long-term immunogenicity and safety of the hepatitis B vaccine HepB-CpG (HEPLISAV-B) compared with HepB-Eng (Engerix-B) in adults with chronic kidney disease. Vaccine. 2023 May 11;41(20):3224-3232. doi: 10.1016/j.vaccine.2023.04.028. Epub 2023 Apr 19. PMID 37085451
- See also: Related Info — http://www.Dynavax.com